CLINICAL TRIAL: NCT05465148
Title: Microbiome Determinants of Neurological and Gastrointestinal Symptoms of Autism Spectrum Disorder (ASD)
Status: Withdrawn | Type: Observational
Why Stopped: Lack of recruitment
Sponsor: Viome (Industry)
Responsible Party: Sponsor
Other Study IDs: V205
Record Dates: First submitted 2022-07-08; First posted 2022-07-19 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Autism Spectrum Disorder
Keywords: Fecal Matter Transplant; FMT; Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ASD: Individuals with Autism Spectrum Disorder indicated by medical records, self diagnosis, or reported by a legally authorized representative. Individuals may be of any age, however, minors (under the age of 18 years) will be required to provide the assent form or a parental permission form, in addition to the Informed Consent Form signed by the parents/guardians prior to any study related activities.

SUMMARY:
This observational study aims to identify human microbiome determinants of the symptoms associate with ASD as well as identify the human microbiome determinants of the success of FMT (fecal matter transplant) therapy and to develop a statistical model that can improve FMT donor-recipient matching. Participants are recruited through NovelBiome only, this study will NOT utilize other clinical sites.

DETAILED DESCRIPTION:
This longitudinal, observational study aims to identify human microbiome determinants of the symptoms associate with ASD as well as identify the human microbiome determinants of the success of FMT therapy and to develop a statistical model that can improve FMT donor-recipient matching.

Participant phenotype data and samples are collected at several time points relative to their receiving FMT therapy.

Participants will collect stool, urine, environmental swabs, saliva, and blood at home via VLS's (Viome Life Sciences) at-home kits mailed to them by VLS. The at-home samples are collected by participants (and when appropriate LAR/guardian). The samples are then returned to VLS via postage-paid mailers (provided). These samples are analyzed by the VLS laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ASD, from medical records, self-diagnosed and/or LAR reported (LAR = legally authorized representative)
* Plans to undergo FMT treatment at a Novel Biome Clinic
* Consented to participate in the study

Exclusion Criteria:

* Active cancer therapy
* Antibiotic use within 30 days prior to starting the FMT therapy. FMT therapy itself starts with antibiotic treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 1000 participants (any biological sex) that have a shipping address within the USA will be enrolled. Participants of all ages will be admitted into the study; minors - under the age of 18 will be required to provide the assent form or a parental permission form, in addition to the Informed Consent Form signed by the parents/guardians prior to any study related activities.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-05-14 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Prevalence of species in samples from people with ASD | 10 years
  Prevalence of species in samples from people with ASD compared to non-ASD samples
Prevalence of species in samples that led to successful FMT therapy | 10 years
  Prevalence of species in samples that led to successful FMT therapy

CONTACTS AND LOCATIONS:
Overall Officials: Momchilo Vuyisich, Principal Investigator — Viome